CLINICAL TRIAL: NCT06128018
Title: A Randomized Trial Comparing Endoscopic UltraSound-guided GasTrojejunostomy (EUS-GJ) and Surgical GastrojejunOstomy (S-GJ) for the Management of Malignant gastRic outlEt Obstruction
Brief Title: Comparing Endoscopic Ultrasound vs Surgical Gastrojejunostomy for Management of GOO.
Acronym: RESTORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2036763
Record Dates: First submitted 2023-10-24; First posted 2023-11-13 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Malignant Gastric Outlet Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-guided gastrojejunostomy (EUS-GJ) (Other): Patients on this arm will undergo the endoscopic procedure.
  Interventions: Procedure: Surgical gastrojejunostomy (S-GJ)
- Surgical gastrojejunostomy (S-GJ) (Other): Patients on this arm will undergo the surgical procedure.
  Interventions: Procedure: EUS-guided gastrojejunostomy (EUS-GJ)

INTERVENTIONS:
Procedure: Surgical gastrojejunostomy (S-GJ) — Surgical gastro-jejunostomy
  Arms: EUS-guided gastrojejunostomy (EUS-GJ)
Procedure: EUS-guided gastrojejunostomy (EUS-GJ) — Endoscopic Ultrasound guided gastro-jejunostomy
  Arms: Surgical gastrojejunostomy (S-GJ)

SUMMARY:
The goal of this interventional study is to learn about the outcomes between two options for the management of malignant gastric outlet obstruction.

DETAILED DESCRIPTION:
The goal of this interventional study is to learn about the outcomes between two options for the management of malignant gastric outlet obstruction. The main question this study aims to answer is:

1. To compare the rates of procedure related adverse events (AE's) between patients undergoing Endoscopy Ultrasound-guided gastro-jejunostomy (EUS-GJ) and Surgical gastro-jejunostomy (S-GJ).

Study participants will be randomized into one of the two standard procedures and followed for up to 12 months post procedure for collection of outcomes related data

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Radiographic OR Endoscopic evidence of an obstructing neoplasm in the distal stomach or duodenum.
3. GOOSS of 0 or 1
4. BOTH surgical and endoscopic GJ are technically and clinically feasible
5. Can understand and is willing to sign informed consent form prior to the initiation of any study procedures (or when applicable the subject's LAR).

Exclusion Criteria:

1. < 18 years of age
2. ECOG >2
3. Expected survival (determined by the treating oncologist) is less than 2 months.
4. Candidates for potential resection of the cancer and obstructed anatomical area (this includes patients with borderline resectable pancreatic cancer)
5. Peritoneal carcinomatosis with associated bowel obstruction on imaging or during laparoscopy
6. Large volume ascites (patients with moderate volume ascites may undergo IR guided drainage prior to randomization)
7. Anatomical factors that technically hinder EUS-GJ OR Surgical-GJ (diffuse tumor involvement in path of LAMS or surgery, surgically altered anatomy that interferes with the ability to perform an anastomosis etc)
8. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Identify safety profile EUS-GJ | 24 Months
  The severity of AEs will be determined using standard American Society of Gastrointestinal Endoscopy (ASGE) Lexicon and AGREE criteria (appendix) in the EUS-GJ group.

SECONDARY OUTCOMES:
Identify safety profile for S-GJ | 24 Months
  The severity of AEs will be determined using Claviden-Dindo classification of surgical complications in the S-GJ group.

CONTACTS AND LOCATIONS:
Overall Officials: Kambiz Kadkhodayan, MD, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Fukami N, Anderson MA, Khan K, Harrison ME, Appalaneni V, Ben-Menachem T, Decker GA, Fanelli RD, Fisher L, Ikenberry SO, Jain R, Jue TL, Krinsky ML, Maple JT, Sharaf RN, Dominitz JA. The role of endoscopy in gastroduodenal obstruction and gastroparesis. Gastrointest Endosc. 2011 Jul;74(1):13-21. doi: 10.1016/j.gie.2010.12.003. No abstract available. PMID 21704805
- [Background] Medina-Franco H, Abarca-Perez L, Espana-Gomez N, Salgado-Nesme N, Ortiz-Lopez LJ, Garcia-Alvarez MN. Morbidity-associated factors after gastrojejunostomy for malignant gastric outlet obstruction. Am Surg. 2007 Sep;73(9):871-5. PMID 17939415
- [Background] Adler DG, Baron TH. Endoscopic palliation of malignant gastric outlet obstruction using self-expanding metal stents: experience in 36 patients. Am J Gastroenterol. 2002 Jan;97(1):72-8. doi: 10.1111/j.1572-0241.2002.05423.x. PMID 11808972
- [Background] Tyberg A, Kumta N, Karia K, Zerbo S, Sharaiha RZ, Kahaleh M. EUS-guided gastrojejunostomy after failed enteral stenting. Gastrointest Endosc. 2015 Apr;81(4):1011-2. doi: 10.1016/j.gie.2014.10.018. Epub 2015 Feb 11. No abstract available. PMID 25680897
- [Background] Khashab MA, Tieu AH, Azola A, Ngamruengphong S, El Zein MH, Kumbhari V. EUS-guided gastrojejunostomy for management of complete gastric outlet obstruction. Gastrointest Endosc. 2015 Oct;82(4):745. doi: 10.1016/j.gie.2015.05.017. Epub 2015 Jun 16. No abstract available. PMID 26092615
- [Background] Itoi T, Ishii K, Tanaka R, Umeda J, Tonozuka R. Current status and perspective of endoscopic ultrasonography-guided gastrojejunostomy: endoscopic ultrasonography-guided double-balloon-occluded gastrojejunostomy (with videos). J Hepatobiliary Pancreat Sci. 2015 Jan;22(1):3-11. doi: 10.1002/jhbp.148. Epub 2014 Aug 24. PMID 25155270
- [Background] Itoi T, Ishii K, Ikeuchi N, Sofuni A, Gotoda T, Moriyasu F, Dhir V, Teoh AY, Binmoeller KF. Prospective evaluation of endoscopic ultrasonography-guided double-balloon-occluded gastrojejunostomy bypass (EPASS) for malignant gastric outlet obstruction. Gut. 2016 Feb;65(2):193-5. doi: 10.1136/gutjnl-2015-310348. Epub 2015 Aug 17. No abstract available. PMID 26282674
- [Background] Binmoeller KF, Shah JN. Endoscopic ultrasound-guided gastroenterostomy using novel tools designed for transluminal therapy: a porcine study. Endoscopy. 2012 May;44(5):499-503. doi: 10.1055/s-0032-1309382. Epub 2012 Apr 24. PMID 22531985
- [Background] Barthet M, Binmoeller KF, Vanbiervliet G, Gonzalez JM, Baron TH, Berdah S. Natural orifice transluminal endoscopic surgery gastroenterostomy with a biflanged lumen-apposing stent: first clinical experience (with videos). Gastrointest Endosc. 2015 Jan;81(1):215-8. doi: 10.1016/j.gie.2014.09.039. PMID 25527056
- [Background] Itoi T, Itokawa F, Uraoka T, Gotoda T, Horii J, Goto O, Moriyasu F, Moon JH, Kitagawa Y, Yahagi N. Novel EUS-guided gastrojejunostomy technique using a new double-balloon enteric tube and lumen-apposing metal stent (with videos). Gastrointest Endosc. 2013 Dec;78(6):934-939. doi: 10.1016/j.gie.2013.09.025. PMID 24237949
- [Background] Khashab MA, Kumbhari V, Grimm IS, Ngamruengphong S, Aguila G, El Zein M, Kalloo AN, Baron TH. EUS-guided gastroenterostomy: the first U.S. clinical experience (with video). Gastrointest Endosc. 2015 Nov;82(5):932-8. doi: 10.1016/j.gie.2015.06.017. Epub 2015 Jul 26. PMID 26215646
- [Background] Tyberg A, Perez-Miranda M, Sanchez-Ocana R, Penas I, de la Serna C, Shah J, Binmoeller K, Gaidhane M, Grimm I, Baron T, Kahaleh M. Endoscopic ultrasound-guided gastrojejunostomy with a lumen-apposing metal stent: a multicenter, international experience. Endosc Int Open. 2016 Mar;4(3):E276-81. doi: 10.1055/s-0042-101789. PMID 27004243